CLINICAL TRIAL: NCT05425927
Title: Validation of 3D Synthetic MRI for Neuroimaging - Prospective, Multicenter, Multireader Investigation
Brief Title: Comparative Study of Conventional MR Images With Synthetically Reconstructed MR Images of the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SyntheticMR (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-003
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Clinical Indication for Brain MRI; Healthy Volunteers
Keywords: neuroimaging

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled from the general imaging population scheduled for an MRI of the brain and healthy volunteers, using the scanner available at the investigational sites. A conventional MRI scan of the brain is taken, and an additional sequence that is processed into synthetic MR images. The conventional and the synthetic MR images from the same subject is compared.
Masking Description: For each subject, conventional and synthetic images will be assessed by blinded, experienced neuroradiologists who will assess the images with regards to radiological findings, image quality, legibility of anatomical structures, and artifacts. The readings will be separated into two reading sessions with a 4-week memory-washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neurologic Synthetic and Conventional MRI (Experimental): MR images of the brain acquired for post-processing with software (SyMRI 15, 3D).
  Comparison is done between the conventional MR images and the post-processed synthetic MR images
  Interventions: Device: SyMRI 15 (3D)

INTERVENTIONS:
Device: SyMRI 15 (3D) — Neurological MRI image collection

SUMMARY:
This study is being conducted for evaluation of 3D Synthetic MRI (SyMRI 15, 3D) for neuroimaging,

DETAILED DESCRIPTION:
This study is a prospective, blinded, multi-center, multi-reader clinical study that is statistically powered for demonstrating non-inferiority of synthetic 3D MR images compared to conventional MR images with respect to sensitivity and specificity of pathological findings.

The study consists of three parts:

* Clinical MR acquisition,
* Synthetic MR post-processing
* Blinded image evaluation of conventional and synthetic images for each subject.

The study will enroll eligible subjects with an already scheduled brain MRI and also healthy volunteers, that meet applicable site MR safety criteria. The routine MRI scan will include approximately 5-20 minutes extra time for the additional images to be taken. This time will be added to the length of the scheduled scan. It is only the time in the MRI scanner that will differ from standard procedures, no other examinations will be performed.

The study consists of one visit, without additional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, aged 0-99 years
* Subject scheduled for MRI of the brain OR Healthy control with passed screening form
* Subject suitable for MRI as judged by investigator
* Subject agrees to 5-20 min extra MRI scan time
* Subject able to understand written and verbal information in English or Spanish
* Provision of informed consent (and assent if applicable)

Exclusion Criteria:

* Have contraindication(s) to MRI scanning per the routine MR Safety Screening policy of the investigational site
* Have severe trauma, disability or pre-existing pathology that is expected to interfere with normal conduct of MRI scanning or complete scanning of the brain
* Have medical condition(s) such as those requiring urgent medical care that, in the opinion of a physician investigator, would prevent safe participation in the study
* Adult subjects (aged 18-99 years) in need of anesthesia during MRI scanning
* Pregnancy at time of enrollment determined according to the clinic's MR Safety Screening policy
* Previous enrollment in this investigation

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Miller, MD, Principal Investigator — Phoenix Children's Hospital
Locations (6):
- United States (6):
  - Phoenix Children's hospital, Phoenix, Arizona
  - ProScan Imaging, Naples, Florida
  - Nemours Children's Health, Nemours Children's Hospital, Florida, Orlando, Florida
  - SimonMed imaging Streeterville, Chicago, Illinois
  - Dent Neurosciences Research Center, New York, New York
  - Diagnostic Imaging Sciences Center (DISC) University of Washington Medical Center (UWMC), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neurological MRI: MR images of the brain acquired for post-processing with software (SyMRI 15, 3D).
  Comparison is done between the conventional MR images and the post-processed synthetic MR images
  SyMRI 15 (3D): Neurological MRI image collection. All participants with complete set of scans that was part of the image review study.
Period: Overall Study
Arm/Group | Neurological MRI
Started | 189
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Neurological MRI Synthetic: MR images of the brain acquired for post-processing with software (SyMRI 15, 3D).
  Comparison is done between the conventional MR images and the post-processed synthetic MR images
  SyMRI 15 (3D): Neurological MRI image collection. All participants with complete set of scans that was part of the image review study.
Arm/Group | Neurological MRI Synthetic
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (23.1)
Age, Customized [Count of Participants; unit: Participants]
  Pediatric (<18 years) | 63
  Adults (>= 18) | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 189
Pathological finding [Count of Participants; unit: Participants] — Based upon the site-determined diagnosis, considered to be the ground truth
  Participants
    Congential malformations | 13
    Infectious/inflammatory/demyelinating | 20
    Intracranial neoplasms | 27
    Toxic and metabolic conditions | 0
    Traumatic lesions | 4
    Vascular disorders of the brain | 26
    Neuro degenerative disorders and hydrocephalus | 13
    Normal/no findings | 86
Anaesthesia used [Count of Participants; unit: Participants]
  Yes | 5
  No | 184

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Pathological Findings (Full Analysis Set)
Description: Sensitivity of pathological findings (true number of participants with pathological findings over assessed number of participants with pathological findings by reader) for synthetic and conventional MR images on the full analysis set. Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: Conventional images and necessary MRI information acquired from participant on exam day (1 day). Synthetic images generated before first reading. Analysis by readers in two readings, first reading: week 0-2, second reading: week 7-8
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Neurologic Synthetic and Conventional MRI: MR images of the brain acquired for post-processing with software (SyMRI 15, 3D).
  Comparison is done between the conventional MR images and the post-processed synthetic MR images
  SyMRI 15 (3D): Neurological MRI image collection. All participants with complete set of scans that was part of the image review study.
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Proportion of participants
  Synthetic | 0.66 [0.59 to 0.74]
  Conventional | 0.68 [0.60 to 0.75]

2. Primary Outcome: Specificity of Pathological Findings (Full Analysis Set)
Description: Specificity of pathological findings (true number of participants with normal/no finding over assessed number of participants with normal/no finding by reader) for synthetic and conventional MR images on the full analysis set. Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Proportion of participants
  Synthetic | 0.85 [0.81 to 0.90]
  Conventional | 0.85 [0.80 to 0.90]

3. Secondary Outcome: Classification of Pathological Findings
Description: Diagnostic accuracy of radiological findings (radiological finding class) for synthetic and conventional MR images on the full analysis set. Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Proportion of participants
  Synthetic | 0.60 [0.55 to 0.65]
  Conventional | 0.60 [0.55 to 0.65]

4. Secondary Outcome: Sensitivity (Adult Population)
Description: Sensitivity of pathological findings (true number of participants with pathological findings over assessed number of participants with pathological findings) for synthetic and conventional MR images in adult population (18-99 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Adult subpopulation 18-99 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 126
Proportion of participants
  Synthetic | 0.68 [0.58 to 0.78]
  Conventional | 0.70 [0.61 to 0.79]

5. Secondary Outcome: Selectivity (Adult Population)
Description: Specificity of pathological findings (true number of participants with normal/no finding over assessed number of participants with normal/no finding) for synthetic and conventional MR images on the in adult population (18-99 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Adult subpopulation 18-99 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 126
Proportion of participants
  Synthetic | 0.84 [0.78 to 0.90]
  Conventional | 0.84 [0.78 to 0.91]

6. Secondary Outcome: Classification of Pathological Findings (Adult Population)
Description: Diagnostic accuracy of radiological findings (radiological finding class) for synthetic and conventional MR images in adult population (18-99 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Adult subpopulation 18-99 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 126
Proportion of participants
  Synthetic | 0.61 [0.55 to 0.68]
  Conventional | 0.61 [0.54 to 0.67]

7. Secondary Outcome: Sensitivity (Pediatric Population)
Description: Sensitivity of pathological findings (true number of participants with pathological findings over assessed number of participants with pathological findings) for synthetic and conventional MR images in pediatric population (0-17 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Pediatric subpopulation 0-17 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 63
Proportion of participants
  Synthetic | 0.64 [0.52 to 0.76]
  Conventional | 0.64 [0.52 to 0.76]

8. Secondary Outcome: Selectivity (Pediatric Population)
Description: Specificity of pathological findings (true number of participants with normal/no finding over assessed number of participants with normal/no finding) for synthetic and conventional MR images on the in pediatric population (0-17 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Pediatric subpopulation 0-17 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 63
Proportion of participants
  Synthetic | 0.90 [0.83 to 0.97]
  Conventional | 0.87 [0.80 to 0.95]

9. Secondary Outcome: Classification of Pathological Findings (Pediatric Population)
Description: Diagnostic accuracy of radiological findings (radiological finding class) for synthetic and conventional MR images in pediatric population (0-17 years). Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The ground truth is the site-determined diagnosis.
Time Frame: as for outcome 1
Population: Pediatric subpopulation 0-17 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 63
Proportion of participants
  Synthetic | 0.57 [0.48 to 0.67]
  Conventional | 0.58 [0.49 to 0.68]

10. Other Pre Specified Outcome: Legibility T1w (Full Analysis Set)
Description: Legibility of anatomical structures, per structure, on the full analysis set for T1w images. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The result for each anatomical structure per image type, independent of reading period, is summarized in corresponding row below.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Number of observations
Units Other Than Participants: Number of observations
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Number analyzed (Number of observations) | 945
Number of observations
  Central sulcus : Synthetic | 940
  Cerebral peduncle : Synthetic | 944
  Cervicomedullary junction : Synthetic | 944
  Head of caudate nucleus : Synthetic | 942
  Middle cerebellar peducle : Synthetic | 944
  Posterior limb of internal capsule : Synthetic | 942
  Central sulcus : Conventional | 938
  Cerebral peduncle : Conventional | 940
  Cervicomedullary junction : Conventional | 944
  Head of caudate nucleus : Conventional | 936
  Middle cerebellar peducle : Conventional | 943
  Posterior limb of internal capsule : Conventional | 933

11. Other Pre Specified Outcome: Legibility T2w (Full Analysis Set)
Description: Legibility of anatomical structures, per structure, on the full analysis set for T2w images. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The result for each anatomical structure per image type, independent of reading period, is summarized in corresponding row below.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Number of observations
Units Other Than Participants: Number of observations
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Number analyzed (Number of observations) | 945
Number of observations
  Central sulcus : Synthetic | 939
  Cerebral peduncle : Synthetic | 942
  Cervicomedullary junction : Synthetic | 943
  Head of caudate nucleus : Synthetic | 934
  Middle cerebellar peducle : Synthetic | 944
  Posterior limb of internal capsule : Synthetic | 937
  Central sulcus : Conventional | 941
  Cerebral peduncle : Conventional | 942
  Cervicomedullary junction : Conventional | 927
  Head of caudate nucleus : Conventional | 923
  Middle cerebellar peducle : Conventional | 942
  Posterior limb of internal capsule : Conventional | 921

12. Other Pre Specified Outcome: Artifacts T1w(Full Analysis Set)
Description: Presence and type of artifacts determined for synthetic T1w images, on the full analysis set determined by all readers. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The result for each artifact per image type, independent of reading period, is summarized in corresponding row below.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Number of observations
Units Other Than Participants: Number of observations
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Number analyzed (Number of observations) | 945
Number of observations
  No artifacts : Synthetic | 851
  Motion artifacts : Synthetic | 29
  In-folding or wrap around artifacts : Synthetic | 1
  Flow or phase-encoding artifacts : Synthetic | 4
  Magic angle effect artifacts : Synthetic | 1
  Water-fat shift/ chemical shift artifacts : Synthetic | 0
  Magnetic susceptibility artifact : Synthetic | 55
  Low resolution : Synthetic | 7
  Low signal to noise : Synthetic | 4
  Low tissue contrast : Synthetic | 5
  No artifacts : Conventional | 820
  Motion artifacts : Conventional | 40
  In-folding or wrap around artifacts : Conventional | 0
  Flow or phase-encoding artifacts : Conventional | 10
  Magic angle effect artifacts : Conventional | 0
  Water-fat shift/ chemical shift artifacts : Conventional | 0
  Magnetic susceptibility artifact : Conventional | 56
  Low resolution : Conventional | 17
  Low signal to noise : Conventional | 22
  Low tissue contrast : Conventional | 21

13. Other Pre Specified Outcome: Artifacts T2w(Full Analysis Set)
Description: Presence and type of artifacts determined for synthetic T2w images, on the full analysis set determined by all readers. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The result for each artifact per image type, independent of reading period, is summarized in corresponding row below.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Number of observations
Units Other Than Participants: Number of observations
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Number analyzed (Number of observations) | 945
Number of observations
  No artifacts : Synthetic | 655
  T2 weighted : Motion artifacts : Synthetic | 33
  In-folding or wrap around artifacts : Synthetic | 1
  Flow or phase-encoding artifacts : Synthetic | 10
  Magic angle effect artifacts : Synthetic | 0
  Water-fat shift/ chemical shift artifacts : Synthetic | 0
  Magnetic susceptibility artifact : Synthetic | 51
  Low resolution : Synthetic | 106
  Low signal to noise : Synthetic | 30
  Low tissue contrast : Synthetic | 164
  No artifacts : Conventional | 600
  Motion artifacts : Conventional | 40
  In-folding or wrap around artifacts : Conventional | 4
  Flow or phase-encoding artifacts : Conventional | 207
  Magic angle effect artifacts : Conventional | 0
  Water-fat shift/ chemical shift artifacts : Conventional | 0
  Magnetic susceptibility artifact : Conventional | 57
  Low resolution : Conventional | 66
  Low signal to noise : Conventional | 64
  Low tissue contrast : Conventional | 56

14. Other Pre Specified Outcome: Inter-rater Agreement (Full Analysis Set)
Description: Inter-rater agreement between all reader's assessment of pathological finding, as well as radiological finding classes, on the full analysis set. Each image was evaluated only once per reader and the agreement is independent of reading session. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The agreement was assessed separately per image type over both reading periods using overall agreement, Fleiss' kappa coefficient, and Gwet's AC1 coefficient. The first reading begun after all image processing was complete.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Proportion of participants
  Pathological finding: Overall agreement (Synthetic) | 0.82 [0.79 to 0.86]
  Pathological finding: Fleiss' kappa coefficient (Synthetic) | 0.64 [0.57 to 0.71]
  Pathological finding: Gwet's AC1 coefficient (Synthetic) | 0.65 [0.58 to 0.72]
  Radiological finding class: Overall agreement (Synthetic) | 0.67 [0.62 to 0.71]
  Radiological finding class: Fleiss' kappa coefficient (Synthetic) | 0.48 [0.42 to 0.53]
  Radiological finding class: Gwet's AC1 coefficient (Synthetic) | 0.63 [0.58 to 0.68]
  Pathological finding: Overall agreement (Conventional) | 0.82 [0.78 to 0.85]
  Pathological finding: Fleiss' kappa coefficient (Conventional) | 0.63 [0.55 to 0.70]
  Pathological finding: Gwet's AC1 coefficient (Conventional) | 0.64 [0.57 to 0.71]
  Radiological finding class: Overall agreement (Conventional) | 0.67 [0.62 to 0.71]
  Radiological finding class: Fleiss' kappa coefficient (Conventional) | 0.48 [0.43 to 0.54]
  Radiological finding class: Gwet's AC1 coefficient (Conventional) | 0.63 [0.58 to 0.68]

15. Other Pre Specified Outcome: Inter-method Agreement (Full Analysis Set)
Description: Inter-method agreement between the different reader's assessment of pathological finding, as well as radiological finding classes, on the full analysis set. Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The agreement was evaluated for all images, independent of reading period and image type, using overall agreement, Fleiss' kappa coefficient, and Gwet's AC1 coefficient. The first reading begun after all image processing was complete.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
Proportion of participants
  Pathological finding: Overall agreement | 0.86 [0.83 to 0.88]
  Pathological finding: Fleiss' kappa coefficient | 0.71 [0.65 to 0.76]
  Pathological finding: Gwet's AC1 coefficient | 0.72 [0.67 to 0.77]
  Radiological finding class: Overall agreement | 0.75 [0.72 to 0.78]
  Radiological finding class: Fleiss' kappa coefficient | 0.61 [0.56 to 0.66]
  Radiological finding class: Gwet's AC1 coefficient | 0.73 [0.69 to 0.76]

16. Other Pre Specified Outcome: Image Quality Score (Full Analysis Set)
Description: Image quality score (1 (Unacceptable) - 5 (Excellent)) per contrast weighting (T1w, T2w) per both image types (conventional and synthetic) where 3,4,5 are deemed acceptable for diagnostic use and 1,2 unacceptable for diagnostic use. Each image was evaluated only once per reader. The images were split between two readings, with a wash-out period of 4 weeks in between. Both readings contained both types of images, synthetic and conventional. The first reading begun after all image processing was complete. The result presented, independent of reading period, is the averaged score per contrast weight and image type with the standard deviation.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
score on a scale
  T1w : Synthetic | 4.6 (0.6)
  T1w : Conventional | 4.5 (0.7)
  T2w : Synthetic | 4.4 (0.7)
  T2w : Conventional | 4.2 (0.8)

17. Other Pre Specified Outcome: Safety (Full Analysis Set)
Description: Incidence of Adverse Events (AE), Adverse Device Effects (ADE), Serious Adverse Events (SAE), Serious Adverse Device Effects (SADE), Unanticipated Adverse Device Effect (UADE), Unanticipated Serious Adverse Device Effect (USADE) and Device Deficiencies (DD). The measurement was assessed in two periods: during exam day after signing consent form (all incidents applicable) and when generating the synthetic images (only device deficiencies) after all exams were performed.
Time Frame: Exam day (1 day), Generation of Synthetic Images (up to 7 weeks)
Measure: Number; unit: events
Arm/Group | Neurologic Synthetic and Conventional MRI
Number analyzed (Participants) | 189
events
  Adverse Events (AE) | 0
  Adverse Device Effects (ADE) | 0
  Serious Adverse Events (SAE) | 0
  Unanticipated Adverse Device Effect (UADE) | 0
  Unanticipated Serious Adverse Device Effect (USADE) | 0
  Device Deficiencies (DD) | 1

ADVERSE EVENTS:
Time Frame: Exam day (1 day), Generation of Synthetic Images (up to 7 weeks)
Arm/Group | Neurologic Synthetic and Conventional MRI
All-Cause Mortality (participants affected / at risk) | 0/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 1/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurologic Synthetic and Conventional MRI (N=189)
Device Deficiencies (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05425927/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05425927/ICF_003.pdf